CLINICAL TRIAL: NCT01882777
Title: ASSESSING THE IMPACT OF WATER FILTERS AND IMPROVED COOK STOVES ON DRINKING WATER QUALITY AND INDOOR AIR POLUTION: A RANDOMISED CONTROLED TRIAL IN RWANDA
Brief Title: Evaluation of a Project to Distribute Water Filters and Cookstoves in Western Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: DelAgua (Other); Portland State University (Other); University of Colorado, Boulder (Other); University of Zurich (Other); Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Thomas Clasen, Dr, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6239
Record Dates: First submitted 2013-02-22; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Faecal Contamination of Household Drinking Water (Environmental Outcome)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Existing water management and cooking practices (No Intervention): Households in the control arm continue following their existing drinking water management and cooking practices
- Provision of water filters and improved cookstoves (Active Comparator): Households in intervention arm are provided with drinking water filters and improved cook stoves
  Interventions: Behavioral: Household drinking water filters and cookstoves

INTERVENTIONS:
Behavioral: Household drinking water filters and cookstoves — The intervention consists of providing households with a household-based drinking water filter (Lifestraw® Family version 2.0) and high efficiency cook stoves (Eco Zoom) as well as instructions on how to use them. The intervention is delivered at community level through community health workers (CHWs). Following initial distribution of the products, CHWs visit households fortnightly to reinforce messages about correct and consistent use.
  Arms: Provision of water filters and improved cookstoves

SUMMARY:
DelAgua Health and Development, Manna Energy and the Rwanda Ministry of Health are collaborating on a project financed by carbon credits that will distribute household-based water filters and high-efficiency cook stoves to approximately 700,000 households in Rwanda. Prior to the full roll out of the campaign, the implementers are conducting a pilot project among 2000 households in western Rwanda. The objectives of this pilot evaluation are to document the delivery of the intervention to the intervention population, assess coverage and uptake of the intervention target households and conduct a 5-month randomised controlled trial among 500 households to assess the impact of the intervention on drinking water quality and indoor air quality.

ELIGIBILITY:
Inclusion Criteria:

* All households in three selected villages

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Thermotolerant coliforms in household drinking water | 5 months
  Faecal contamination levels (thermotolerant coliforms) in household drinking water. Household drinking water quality will be monitored monthly over a 5-month period.

SECONDARY OUTCOMES:
Particulate matters 2.5 mg/m3 (PM2.5) concentrations | once
  PM2.5 concentrations measured in reported main cooking area once (24-hour period) in a sub-sample of 120 households.
Adherence - use of water filters and cookstoves | 5 months
  Questionnaires, direct observations and electronic monitoring devices

CONTACTS AND LOCATIONS:
Locations (1):
- Manna Energy Ltd., Kigali, Rwanda

REFERENCES:
- [Derived] Rosa G, Majorin F, Boisson S, Barstow C, Johnson M, Kirby M, Ngabo F, Thomas E, Clasen T. Assessing the impact of water filters and improved cook stoves on drinking water quality and household air pollution: a randomised controlled trial in Rwanda. PLoS One. 2014 Mar 10;9(3):e91011. doi: 10.1371/journal.pone.0091011. eCollection 2014. PMID 24614750